CLINICAL TRIAL: NCT01317108
Title: Adjuvant Chemotherapy in Node-negative Breast Cancer: Chemo N0
Brief Title: Prognostic and Predictive Impact of uPA/PAI-1
Acronym: ChemoN0
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ChemoN0; GR280/4 (Other Grant/Funding Number: German Research Association)
Record Dates: First submitted 2011-02-21; First posted 2011-03-17 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: node-negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (No Intervention): Low uPA/PAI-1: Observation
- B2 (No Intervention): High uPA/PAI-1: Observation
- B3 (No Intervention): High uPA/PAI-1: refused randomization
- B1 (Active Comparator): High uPA/PAi-1: CMF chemotherapy
  Interventions: Drug: CMF Chemotherapy

INTERVENTIONS:
Drug: CMF Chemotherapy
  Arms: B1

SUMMARY:
Chemo-N0 (1993-1998) is the first prospective randomized multicenter trial in N0 BC designed to prospectively evaluate the clinical utility of a biomarker. It used uPA/PAI 1 as stratification criteria and randomized high-risk patients to chemotherapy versus observation; low-risk patients remained without any systemic therapy. The trial was designed to answer two principle questions:

1. Can the reported prognostic impact of uPA and PAI 1 be validated in a prospective multicenter therapy trial? Does low uPA/PAI 1 identify those low-risk N0 patients who are candidates for being spared necessity and burden of adjuvant chemotherapy?
2. Do uPA/PAI 1 high-risk patients benefit from adjuvant CMF chemotherapy?

ELIGIBILITY:
Inclusion Criteria:

* N0 breast cancer patients tumor size >/= 1 and </= 5 cm in diameter undergoing standard loco-regional treatment

Exclusion Criteria:

* M1 status

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 1993-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Prognostic impact of uPA/PAI-1: Number of patients disease-free in low vs. high risk groups according to uPA/PAI-1 | DFS at 3, 5, and 10 years (depending on analysis time point)
  Interim analyses planned at 4.5, 6.5, and 8.5 years after first patient in. Final analysis scheduled at 10.5 years after last patient in.
The benefit of adjuvant chemotherapy in high-risk group according to uPA/PAI-1: Number of patients disease-free vs. those relapsed at the given time points | DFS at 3, 5, and 10 years (depending on analysis time point)
  Interim analyses planned at 4.5, 6.5, and 8.5 years after first patient in. Final analysis scheduled at 10.5 years after last patient in.

SECONDARY OUTCOMES:
Overall survival | at 3, 5, and 10 years (depending on analysis time point).
  Interim analyses planned at 4.5, 6.5, and 8.5 years after first patient in. Final analysis scheduled at 10.5 years after last patient in.

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Jaenicke, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf

REFERENCES:
- [Result] Janicke F, Prechtl A, Thomssen C, Harbeck N, Meisner C, Untch M, Sweep CG, Selbmann HK, Graeff H, Schmitt M; German N0 Study Group. Randomized adjuvant chemotherapy trial in high-risk, lymph node-negative breast cancer patients identified by urokinase-type plasminogen activator and plasminogen activator inhibitor type 1. J Natl Cancer Inst. 2001 Jun 20;93(12):913-20. doi: 10.1093/jnci/93.12.913. PMID 11416112
- [Derived] Harbeck N, Schmitt M, Meisner C, Friedel C, Untch M, Schmidt M, Sweep CG, Lisboa BW, Lux MP, Beck T, Hasmuller S, Kiechle M, Janicke F, Thomssen C; Chemo-N 0 Study Group. Ten-year analysis of the prospective multicentre Chemo-N0 trial validates American Society of Clinical Oncology (ASCO)-recommended biomarkers uPA and PAI-1 for therapy decision making in node-negative breast cancer patients. Eur J Cancer. 2013 May;49(8):1825-35. doi: 10.1016/j.ejca.2013.01.007. Epub 2013 Mar 13. PMID 23490655